CLINICAL TRIAL: NCT02915406
Title: cliniMACs HUD for T Cell Depletion
Status: No longer available | Type: Expanded Access
Sponsor: University of Miami (Other)
Collaborators: Jackson Health System (Other)
Responsible Party: Principal Investigator, Gary Kleiner, Associate Professor of Pediatrics, University of Miami
Other Study IDs: 20160472
Record Dates: First submitted 2016-09-23; First posted 2016-09-27 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: x Linked Combined Immunodeficiency
MeSH Terms: conditions — X-Linked Combined Immunodeficiency Diseases

INTERVENTIONS:
Device: CliniMACs

SUMMARY:
This protocol is designed to enable access to related or unrelated CD34 cells manufactured using the CliniMACS (Miltenyi) under the HUD designation for patients needing T cell depleted allogeneic grafts for hematopoietic stem cell transplant (HSCT). This will include patients with inherited immunodeficiency disorders as well as patients with malignancies, bone marrow failure, and other rare diseases amenable to HSCT. Finally, patients with poor graft function and Graft Versus Host Disease(GVHD) after a previous HSCT may require a boost of T-cell depleted donor Peripheral Blood Stem Cell (PBSCs) or bone marrow cells that are CD34 selected using the CliniMACS device ENROLLMENT BY INVITATION ONLY

ELIGIBILITY:
Inclusion Criteria:

severe combined immune deficiency need for stem cell boost

Exclusion Criteria:

n/a

Max Age: 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Gary Kleiner, MDPhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States